CLINICAL TRIAL: NCT06744608
Title: Effectiveness of Structured Myofascial Release in the Treatment of Primary Dysmenorrhea
Brief Title: Effectiveness of Structured Myofascial Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Buse Sert, MSc physiotherapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDIPOLU-FTR-BS-01
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Primary Dysmenorrhea
Keywords: Myofascial Release; TENS (transcutaneous electrical nerve stimulation)
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: 1. Structured myofascial release group
  2. Tens (transcutaneous electrical nerve stimulation) group
  3. group that includes lifestyle changes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Structured Myofascial Release (Active Comparator): The treatment program consisting of myofascial release techniques includes the following applications; 1. Anterolateral abdominal wall release (Until relaxation is felt); Along the fundus of the uterus, along the ovaries and the broad ligament of the uterus, combined mobilization with rotation of the uterus and hips in the supine position and sacral mobilization for three minutes. Myofascial release was started by placing the fingers/dorsal side of the hand on the fascia. Pressure was applied on the soft tissue. After the restricted layer was felt, the fascia was moved along the surface while in contact with the lower layers. The technique was applied for an average of 60-90 seconds, but if necessary, it was continued until relaxation was felt.
  Interventions: Other: Structured Myofascial Release
- TENS (transcutaneous electrical nerve stimulation) (Active Comparator): The TENS (transcutaneous electrical nerve stimulation) treatment program was applied by a physiotherapist using two 50X50 mm electrodes on the lower abdomen using conventional TENS at 200 μs, 100 Hz, and 30 min.
  .
  Interventions: Device: tens (transcutaneous electrical nerve stimulation)
- lifestyle changes (Active Comparator): Within the scope of education including lifestyle changes; Good nutrition. (what to take and what to avoid), supplements, relaxation training, meditation, exercise recommendations, avoiding tobacco smoke, warm showers, quality sleep (at least 6-8 hours), wearing comfortable clothes are included in the recommendations.
  Interventions: Behavioral: lifestyle changes

INTERVENTIONS:
Other: Structured Myofascial Release — haftada 2 seans 8 hafta boyunca toplam 16 seans uygulama yapıldı
  Arms: Structured Myofascial Release
Device: tens (transcutaneous electrical nerve stimulation) — A total of 16 sessions of application were applied to the groups, 2 sessions per week for 8 weeks.
  Arms: TENS (transcutaneous electrical nerve stimulation)
Behavioral: lifestyle changes — A presentation including lifestyle changes was prepared and training was provided.
  Arms: lifestyle changes

SUMMARY:
The aim of our research is to examine the effects of myofascial release techniques on symptoms in patients with primary dysmenorrhea. With this research, we aim to improve the clinical symptoms, pain and tension of primary dysmenorrhea with a structured manual therapy consisting of myofascial release and sacral mobilization in individuals with primary dysmenorrhea and an educational program that includes changes in daily life. Can Structured Myofascial Release Techniques Reduce Pain and Other Symptoms in Primary Dysmenorrhea? H0: Myofascial release techniques applied to individuals with primary dysmenorrhea have no effect on symptoms. H1: Myofascial release techniques applied to individuals with primary dysmenorrhea have an effect on symptoms.

DETAILED DESCRIPTION:
Although primary dysmenorrhea is a common problem, especially among young women, there is generally no approach aimed at solving the main issue apart from symptomatic treatment or medication. Due to the side effects of medical treatments, many patients tend to opt for cheaper, non-medical, and non-aggressive methods.

The Weissman scale is scored between 0 and 3, where:

0: No dysmenorrhea

1. Minimal (Able to work but feels discomfort)
2. Moderate (Able to work but feels significant discomfort)
3. Severe (Unable to work, bedridden) According to the Weissman scale, women in groups 1 and 2 continue with their daily lives or work/school but experience significant declines in their quality of life. On the other hand, individuals in group 3 suffer from work loss. Primary dysmenorrhea is associated with a significant economic burden caused by absenteeism and 2 to 3 times higher healthcare costs. Considering this cycle repeats in every menstrual period, a treatment approach is needed not only to alleviate symptoms but also to address the pathophysiological mechanisms of dysmenorrhea. The aim is to reduce elevated prostaglandin levels, decrease increased uterine contractions, relieve ischemia, and improve blood flow using structured myofascial release techniques.

Structured Myofascial Release Techniques

Myofascial release techniques involve manual physiotherapy administered by a physiotherapist to eliminate myofascial trigger points, reduce muscle tension, and alleviate associated pain. Structured myofascial release techniques aim to:

Provide relaxation in smooth muscles and ligaments through direct techniques to reduce increased uterine contractions.

Achieve neural relaxation via sacral mobilization. Incorporate a dual relaxation protocol involving both mechanical correction and stimulation of the parasympathetic nervous system.

It is thought that applying these two methods together increases the likelihood of treatment success. In 2022, a study demonstrated that myofascial release provided more effective relaxation and symptom reduction compared to pelvic floor exercises in patients with primary dysmenorrhea. This project aims to evaluate the effectiveness of myofascial release techniques and investigate whether the treatment effect persists after the intervention.

TENS (transcutaneous electrical nerve stimulation)

In the TENS group, pain is reduced by direct application to the lower abdominal area through the gate control theory. TENS is hypothesized to have two effects:

Elevating the threshold of pain signals caused by uterine hypoxia and hypercontractility by sending afferent impulses via the large-diameter sensory fibers of the same nerve root, thereby reducing the perception of painful uterine signals.

Stimulating endorphin release from peripheral nerves and the spinal cord Research Question and Hypotheses Research Question: Can structured myofascial release techniques reduce pain and other symptoms in the treatment of primary dysmenorrhea?

H0: Myofascial release techniques have no effect on the symptoms of individuals with primary dysmenorrhea.

H1: Myofascial release techniques have an effect on the symptoms of individuals with primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Primary dysmenorrhea diagnosed by a specialist gynecologist with 'Ultrasonography',
* Complaints of pain and spasm in the first 2 days of the menstrual cycle,
* Being two or above on the Weissmann scale,
* Being between the ages of 18-30,
* Volunteering to participate in the study

Exclusion Criteria:

* Having pelvic pathology,
* Having a history of previous pregnancy,
* Using a medication that causes or affects dysmenorrhea,
* Being pregnant,
* Using intrauterine or oral contraceptives,
* Having a Body Mass Index (BMI) of 30 and above

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 41 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
McGILL Pain Scale Short Form | three mounth
  The McGill pain questionnaire consists of four sections. In the first section, the individual marks the location of the pain on the body diagram and determines whether the pain comes from deep or superficial. In the second section, there are 20 word groups that examine pain in terms of sensory, perceptual and evaluative aspects. The individual is asked to select a set of words that fit their pain and mark the word that fits their pain within the selected set. The third section includes the relationship between pain and time. In the fourth section, five word groups ranging from "mild" pain to "unbearable" pain are defined to determine the severity of pain. The McGill Pain Questionnaire determines the location of the pain, the feeling it creates in the individual, its relationship with time, its severity and the level of pain that can be experienced by the individual. A high score indicates high level pain.

SECONDARY OUTCOMES:
Menstruation Symptom Scale | three mounth
  Menstrual Symptom Questionnaire (MSQ): The MSQ is a five-point Likert-type scale consisting of twenty-two items. Participants are asked to rate the symptoms they experience related to menstruation between 1 (never) and 5 (always). The scale has three sub-dimensions: 'Negative Effects/Somatic Complaints' (Items 1-13), 'Menstrual Pain Symptoms' (Items 14-19) and 'Coping Methods' (Items 20-22). The highest score that can be obtained from the scale is 110, and the lowest score is 22. The MSQ score is calculated by taking the total score average of the items in the scale. An increase in the score average indicates an increase in the severity of menstrual symptoms.
Functional and Emotional Dysmenorrhea Scale | three mounth
  This is a 14-item Likert-type scale used to measure dysmenorrhea functionally and emotionally. The options on the scale are: (1) It is not like my situation at all, (2) It is not like my situation at all, (3) It is both similar and not like my situation, (4) It is considered similar to my situation, (5) It is very similar to my situation. There are no reverse items in the scale items. The scale was developed to provide functional and emotional measurement of dysmenorrhea. As the scores obtained from the scale increase, the functional and emotional effects of dysmenorrhea also increase.
Myotonometry (MyotonPRO) | three mounth
  Myotonometry is an objective measurement method for measuring the physiological properties of muscle tone, including stiffness. MyotonPRO is a small, non-invasive, handheld myotonometer that provides an objective measurement of the mechanical properties of muscles in vivo. This measurement is a non-invasive approach, where the response of the muscle is recorded using small mechanical stimuli given by the device. In our case, the measurement will be performed in the lower abdomen, at the level of the uterine fundus.

CONTACTS AND LOCATIONS:
Overall Officials: SERT BUSE, Principal Investigator — İstanbul Medipol University
Locations (1):
- Tepe Medical Center, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No